CLINICAL TRIAL: NCT02267369
Title: The Causal Impact of Online Social Media on Physical Activity: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 819455
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Physical Activity
Keywords: online; social media; online social network; physical activity; message
MeSH Terms: conditions — Motor Activity | interventions — Social Conditions

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Basic fitness program (Active Comparator): The control condition provides study participants with online tools for enrolling in offline fitness workshops offered by the university's recreation department and recording their progress in the program. All fitness workshops are pre-programmed in an online calendar. Upon clicking a workshop, participants can read a detailed description and register for it directly on the calendar. The registration then triggers a confirmation email sent to the participant immediately and a reminder email 12 hours before the workshop starts. In addition, an online tracking tool is built that participants can use to keep a daily journal of their health activities and fitness status.
  Interventions: Behavioral: Basic fitness program
- Media-assisted fitness program (Experimental): The media condition evaluates the effects of informational and motivational messages on physical activity by supplementing the basic program tools with promotional media, including: "high arousal" videos encouraging physical activity, real-time email notifications about upcoming fitness workshops, and informational graphics with exercise tips and motivational messages. In the media condition, participants receive two videos on the website and one informational graphic that encourage physical activity on a weekly basis.
  Interventions: Behavioral: Media-assisted fitness program
- Social network-assisted fitness program (Experimental): The social condition, by contrast, omits the media content. Instead, the basic program is supplemented with a network of four to six anonymous "health peers," composed of other participants of the program. Within the program website, each participant is able to see their peers' basic profile information, as well as information about their peers' progress in the program, and real-time notifications about their peers' completion of program activities. These networks do not provide any added incentives or additional content to promote physical activity, nor can participants directly communicate with, or "message" their peers through the website.
  Interventions: Behavioral: Social network-assisted fitness program

INTERVENTIONS:
Behavioral: Media-assisted fitness program — Participants can register workshops online, track program participation, and receive promotional health messages online.
  Other Names: Media condition
  Arms: Media-assisted fitness program
Behavioral: Social network-assisted fitness program — Participants can register workshops online and track program participation. Participants are put into anonymous online social networks and receive real-time activity updates from 4-6 peers.
  Other Names: Social condition
  Arms: Social network-assisted fitness program
Behavioral: Basic fitness program — Participants can register workshops online and track program participation.
  Other Names: Control condition
  Arms: Basic fitness program

SUMMARY:
The overall objective of this research is to collect data for understanding whether messages in online environments impact fitness attitudes and behaviors. In particular, the study aims to experimentally examine what features of online social media - promotional messaging or peer networks - impact offline fitness measures (such fitness workshop enrollment and self-reported physical activity level). The study partners with an existing fitness program at a large northeastern university, which provides a 13-week fitness program for graduate and professional students at the university. The program begins with a university-run eligibility assessment of specific fitness measures for all participants, who win prizes for improvements in program participation and health behavior outcomes. The fitness program consists of semester-long series of workshops offered through the university's recreation department. The randomized trial constructs an online social media platform for the fitness program that provides a way to send either promotion health messages or messages about peer activities to the online community.

DETAILED DESCRIPTION:
Sedentary lifestyle among university students and young adults has become a global epidemic. Widespread use of social media is both a contributing factor, and a potential solution; however the cost-effective use of social media to promote fitness on college campuses is poorly understood. This study aims to identify what features of social media - promotional messaging or peer networks - can increase physical activity levels.

In this randomized controlled trial, participants are randomized to three conditions: basic online program for enrolling in university-run weekly fitness workshops, media condition that supplements the basic program with promotional media messages, and a social condition that replaces the media content with a network of peers. Participants are limited to graduate and professional students at a large northeastern university.

ELIGIBILITY:
Inclusion Criteria:

* Graduate and professional students at a large northeastern university.
* Logging in to the study website at least once after online registration

Exclusion Criteria:

* Inability to perform physical activities (e.g., broken limbs), and underlying diseases that were likely to affect participant safety. Ineligibility is determined by the Department of Recreation and Health Services at the university.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Fitness workshop enrollment | Up to 3 months
  Participants' enrollment in fitness workshops is recorded when participants digitally confirm their workshop registration. Workshop instructors confirm the attendance of enrolled participants. Enrollment is assessed up to 3 months from date of randomization.

SECONDARY OUTCOMES:
Change from baseline in participants' self-reported physical activity level | Baseline and 3 months
  At the baseline and post-program (3 months) online surveys, participants answer the question: "On how many of the past 7 days did you participate in physical activity for at least 30 minutes that did not make you sweat or breathe hard, such as fast walking, slow bicycling, and skating?" Responses to the question range from 0 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Damon M. Centola, Ph.D, Principal Investigator — Annenberg School for Communication, University of Pennsylvania

REFERENCES:
- [Background] Valle CG, Tate DF, Mayer DK, Allicock M, Cai J. A randomized trial of a Facebook-based physical activity intervention for young adult cancer survivors. J Cancer Surviv. 2013 Sep;7(3):355-68. doi: 10.1007/s11764-013-0279-5. Epub 2013 Mar 27. PMID 23532799
- [Background] Cavallo DN, Tate DF, Ries AV, Brown JD, DeVellis RF, Ammerman AS. A social media-based physical activity intervention: a randomized controlled trial. Am J Prev Med. 2012 Nov;43(5):527-32. doi: 10.1016/j.amepre.2012.07.019. PMID 23079176
- [Background] Cobb NK, Graham AL. Health behavior interventions in the age of facebook. Am J Prev Med. 2012 Nov;43(5):571-2. doi: 10.1016/j.amepre.2012.08.001. No abstract available. PMID 23079184
- [Background] Eysenbach G, Powell J, Englesakis M, Rizo C, Stern A. Health related virtual communities and electronic support groups: systematic review of the effects of online peer to peer interactions. BMJ. 2004 May 15;328(7449):1166. doi: 10.1136/bmj.328.7449.1166. PMID 15142921
- [Background] Centola D. The spread of behavior in an online social network experiment. Science. 2010 Sep 3;329(5996):1194-7. doi: 10.1126/science.1185231. PMID 20813952
- [Background] Centola D. An experimental study of homophily in the adoption of health behavior. Science. 2011 Dec 2;334(6060):1269-72. doi: 10.1126/science.1207055. PMID 22144624
- [Background] Korda H, Itani Z. Harnessing social media for health promotion and behavior change. Health Promot Pract. 2013 Jan;14(1):15-23. doi: 10.1177/1524839911405850. Epub 2011 May 10. PMID 21558472
- [Background] Bennett GG, Glasgow RE. The delivery of public health interventions via the Internet: actualizing their potential. Annu Rev Public Health. 2009;30:273-92. doi: 10.1146/annurev.publhealth.031308.100235. PMID 19296777
- [Background] Strecher V. Internet methods for delivering behavioral and health-related interventions (eHealth). Annu Rev Clin Psychol. 2007;3:53-76. doi: 10.1146/annurev.clinpsy.3.022806.091428. PMID 17716048
- [Derived] Zhang J, Brackbill D, Yang S, Centola D. Efficacy and causal mechanism of an online social media intervention to increase physical activity: Results of a randomized controlled trial. Prev Med Rep. 2015 Aug 13;2:651-7. doi: 10.1016/j.pmedr.2015.08.005. eCollection 2015. PMID 26844132